CLINICAL TRIAL: NCT01794221
Title: The Role of 2-octyl Cyanoacrylate in Prevention of Recurrent Adhesions After Circumcision
Acronym: Circglue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1290443
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Phimosis; Adhesions
Keywords: circumcision; 2 octyl cyanoacrylate; phimosis
MeSH Terms: conditions — Phimosis; Tissue Adhesions | interventions — Surgical Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stitches only (Active Comparator): Stitches only closing circumcision wound
  Interventions: Procedure: stitches only
- Stitches and skin adhesive (Experimental): application of 2-octyl cyanoacrylate skin adhesive.
  Interventions: Procedure: stitches and skin adhesive

INTERVENTIONS:
Procedure: stitches and skin adhesive — In addition to stitches, 2-octyl cyanoacrylate skin adhesive will be applied to the circumcision wound.
  Other Names: skin adhesive
  Arms: Stitches and skin adhesive
Procedure: stitches only — standard of care
  Arms: Stitches only

SUMMARY:
The objective of this study is to evaluate whether 2-octyl cyanoacrylate skin adhesive decreased the incidence of recurrent adhesions after circumcision. The investigators hypothesize that the incidence of recurrent adhesions will be decreased with use of 2-octyl cyanoacrylate skin adhesive.

DETAILED DESCRIPTION:
The objective of this study is to evaluate whether 2-octyl cyanoacrylate skin adhesive decreased the incidence of recurrent adhesions after circumcision. The investigators hypothesize that the incidence of recurrent adhesions will be decreased with use of 2-octyl cyanoacrylate skin adhesive.

Secondary Objective(s) To assess parent satisfaction and comfort level after circumcision with use of 2-octyl cyanoacrylate skin adhesive and compare to those undergoing circumcision without the use of 2-octyl cyanoacrylate skin adhesive.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing circumcision
* Only male patients under the age of 7 years will be eligible

Exclusion Criteria:

* Any patient over 7 years of age
* Previous circumcision
* Any parents who are not English language speaking

Ages: 1 Day to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 422 (Actual)
Dates: Start 2012-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Post circumcision adhesions | 3-6 weeks
  Evaluation for adhesions

SECONDARY OUTCOMES:
Parent satisfaction and comfort level with circumcision results | 3-6 weeks
  Parent survey at follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No